CLINICAL TRIAL: NCT00806546
Title: An Open-Label Study to Evaluate the Safety of NP101, a Sumatriptan Iontophoretic Transdermal Patch, in the Treatment of Acute Migraine Over 12 Months
Brief Title: An Open-Label Study to Evaluate the Safety of NP101 in the Treatment of Acute Migraine Over Twelve Months
Acronym: NP101-009
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NuPathe Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROT-15-NP101-009
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2013-03-20 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NP101 (Experimental): sumatriptan iontophoretic transdermal patch
  Interventions: Drug: NP101

INTERVENTIONS:
Drug: NP101 — NP101 study patch four hour application

SUMMARY:
This study will use an open-label design to evaluate the safety of NP101. Adult subjects who meet the enrollment criteria will be treated with NP101 (sumatriptan succinate iontophoretic transdermal patch) for acute migraine attacks over a 12 month period.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult male or female, age range 18 years to 65 years.
* Subject has a diagnosis of migraine headache, with or without aura, as defined in the ICHD-II and the diagnosis was made before the age of 50.
* Subject experiences mild to severe headaches during a migraine attack based on subject testimony.
* Subject has at least a one year history of migraine based upon subject testimony.
* Subject typically experiences at least two migraine headaches per month based on subject testimony.
* Subject will be judged to be in good health, based upon the results of a medical history, physical examination, vital signs, ECG and laboratory profile. Subjects will not have any clinically significant abnormal laboratory parameters, vital signs or ECG parameters in order to qualify for enrollment.
* Female subject of childbearing potential (not surgically sterile or 2 years postmenopausal) must have a negative pregnancy test at screening and prior to enrollment.
* Subject must have a negative drug screen.
* Subject must be capable of reading and understanding either English or Spanish subject information materials. Be able to successfully apply a practice patch, carry-out all subject procedures, and be able to voluntarily sign and date an IC agreement approved by an IRB.
* Subject has at least two acceptable patch application sites (upper arms or upper thighs) that are relatively hair free and has no scars, tattoos, scratches or bruises.
* In the investigator's opinion the subject is on a stable medication regimen.

Exclusion Criteria:

* Subject has more than 15 headache days per month for any of the three months prior to screening.
* Subject has suspected or confirmed cardiovascular disease that contraindicates study participation.
* Subject has a history of epilepsy or condition associated with a lowered seizure threshold.
* Subject has Raynaud's disease.
* Subject has a history of basilar or hemiplegic migraines.
* Subject has a history (within 1 year) or current evidence of drug or alcohol abuse or dependence.
* Subject has taken non-triptan serotonergic drugs including SSRIs (including Wellbutrin), SNRIs, TCAs, MAOIs or preparations containing St. John's Wort within 1 month prior to screening and/or is planning to start any of these medications during the study.
* Subject is unwilling to discontinue use of a PD5 inhibitor (e.g. Viagra®, Levitra®, or Cialis®) through the Final Visit.
* Subject has a history of a significant allergy or hypersensitivity to any component of the study patch used in this study.
* Subject has any generalized skin irritation or disease including eczema, psoriasis, melanoma, or contact dermatitis that would affect transdermal absorption of sumatriptan and / or affect the subjects ability to assess skin irritation.
* Subject has clinically significant abnormal laboratory parameters, vital signs or ECG parameters.
* Subject is known to be hepatitis B, hepatitis C or HIV positive.
* Subject has a diagnosis of bipolar disorder or current major depressive disorder, or has any other medical or psychiatric condition, that in the investigator's opinion would make the subject unsuitable for enrollment / participation in the study.
* Subject has hepatic dysfunction defined as SGOT/AST or SGPT/ALT ≥ 2 times the upper limit of normal (ULN) range, or alkaline phosphatase or total bilirubin ≥ 1.5 times the ULN range or if in the opinion of the Investigator the subject's history, physical examination or other laboratory tests suggest hepatic dysfunction.
* Female subject who is pregnant, breast feeding, or if of childbearing potential, is not using or is unwilling to use an effective form of contraception during the study and for a period of 30 days following dosing.
* Subject has known history of failure to respond to sumatriptan (ineffective or poorly tolerated).
* Subject has participated in a clinical study within 30 days of screening or is planning to participate in another clinical study.
* Subject has been previously enrolled in NP101-008.
* Subject is electrically sensitive (e.g., prior iontophoresis with adverse outcome related to the current delivered by the device) or who have electrically sensitive support systems (e.g., pacemaker) or other medical condition that in the investigator's opinion would make the subject unsuitable for enrollment in the study.
* Subject who is considered by investigator or NuPathe, for any reason, to be an unsuitable candidate for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pierce, M.D., PhD., Study Director — NuPathe Inc.
Locations (31):
- United States (31):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Irvine, California
  - Newport Beach, California
  - San Francisco, California
  - Santa Monica, California
  - Walnut Creek, California
  - Fairfield, Connecticut
  - Hallandale, Florida
  - Ocala, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Savannah, Georgia
  - Crestview Hills, Kentucky
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Mount Vernon, New York
  - Plainview, New York
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Clarksville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Alexandria, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated March 2009 and completed in May 2011. Patients were enrolled from 34 investigative sites across the United States.
Groups:
- NP101: The NP101 patch contained 86 mg of sumatriptan and was designed to deliver approximately 6.5 mg of sumatriptan over 4 hours. Patients were asked to use study patches to treat migraine episodes with mild to severe headache pain for up to 12 months, during which they were permitted to apply (to the upper arms or thighs) a maximum of 6 patches within a 30-day period.
Period: Overall Study
Arm/Group | NP101
Started | 514 (35 subjects were enrolled but did not treat for a total of 479 subjects in the safety population)
Completed | 207
Not Completed | 307
Not completed — Enrolled, not treated | 35
Not completed — Lost to Follow-up | 32
Not completed — Adverse Event | 74
Not completed — Withdrawal by Subject | 75
Not completed — Protocol Violation | 49
Not completed — Various | 42

BASELINE CHARACTERISTICS:
Population: Patients were asked to use study patches to treat migraine episodes with mild to severe headache pain for up to 12 months. The safety population included all subjects who applied at least one NP101 patch. Of the 514 subjects enrolled, 35 subjects did not treat for a total of 479 subjects in the safety population.
Arm/Group | NP101
Number analyzed (Participants) | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 479
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 392
  Male | 87
Region of Enrollment [Number; unit: participants]
  United States | 479

OUTCOME MEASURES:

1. Primary Outcome: Subject Self-examination of Skin Irritation
Description: For each patch application, subjects performed a self-examination of skin irritation using a 5-point scale (0=no redness; 1=minimal skin redness; 2=moderate skin redness with sharp borders; 3=intense skin redness with or without swelling; 4=intense skin redness with blisters or broken skin).
Time Frame: 24 hours post patch application
Population: Per protocol, all subjects who applied at least one NP101 study patch were included in the safety population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Patches
Arm/Group | NP101
Number analyzed (Participants) | 479
Number analyzed (Patches) | 7395
scores on a scale | 0.6 (0.86)

ADVERSE EVENTS:
Time Frame: All adverse events were collected from Screening until 30 days after the last study visit.
Arm/Group | NP101
Serious Adverse Events (participants affected / at risk) | 9/479
Other Adverse Events (participants affected / at risk) | 177/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NP101 (N=479)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Goiter (Endocrine disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NP101 (N=479)
Application site discoloration (General disorders) | 28 (28)
Application site dryness (General disorders) | 27 (27)
Application site pain (General disorders) | 93 (93)
Application site paraesthesia (General disorders) | 26 (26)
Application site pruritus (General disorders) | 67 (67)
Application site reaction (General disorders) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the study agreement, Investigators shall have the right to publish or present information and/or data arising from the study, provided the text of any such publication or presentation is submitted for review at least thirty days prior to submission for publication or other disclosure and NuPathe shall have the right to request the removal of any confidential information